CLINICAL TRIAL: NCT00924989
Title: A Randomized, Double-blind, Placebo-controlled, Phase 3 Study of OSI-906 in Patients With Locally Advanced or Metastatic Adrenocortical Carcinoma
Brief Title: A Study of OSI-906 in Patients With Locally Advanced or Metastatic Adrenocortical Carcinoma
Acronym: GALACCTIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OSI-906-301; 2009-012820-97 (EudraCT Number)
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Adrenocortical Carcinoma
Keywords: Adrenocortical carcinoma; OSI-906; ACC; GALACCTIC; Insulin-like growth factor-1 receptor (IGF-1R)
MeSH Terms: conditions — Adrenocortical Carcinoma; Insulin-Like Growth Factor I, Resistance To | interventions — 3-(8-amino-1-(2-phenylquinolin-7-yl)imidazo(1,5-a)pyrazin-3-yl)-1-methylcyclobutanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: OSI-906 (Experimental): 150 mg twice daily
  Interventions: Drug: OSI-906
- Arm B: Placebo (Placebo Comparator): Matching placebo twice daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: OSI-906 — Administered orally
  Other Names: linsitinib
  Arms: Arm A: OSI-906
Other: Placebo — Matching placebo administered orally
  Arms: Arm B: Placebo

SUMMARY:
A multicenter, randomized, double-blind, placebo-controlled, phase 3 study of single-agent OSI-906 in patients with locally advanced/metastatic Adrenocortical Carcinoma (ACC) who received at least 1 but no more than 2 prior drug regimens

DETAILED DESCRIPTION:
Patients will be randomized 2:1 to receive either single agent OSI-906 (Arm A) or placebo (Arm B) and will be stratified according to prior systemic cytotoxic chemotherapy for ACC, and Eastern Cooperative Oncology Group (ECOG) performance status, and use of >= 1 oral antihyperglycemic therapy at randomization

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adrenocortical carcinoma that is locally advanced or metastatic and not amenable to surgical resection.
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (RECIST) (version 1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) <= 2
* Predicted life expectancy >= 12 weeks.
* At least 1 but no more than 2 prior drug regimens (including molecular targeted therapy, systemic cytotoxic chemotherapy, biologics, and/or vaccines) for locally advanced/metastatic ACC.
* A minimum of 3 weeks must have elapsed between the end of prior treatment and randomization.
* All patients must have received prior mitotane, either as neoadjuvant, adjuvant, or locally advanced/metastatic therapy.
* Adjuvant and neoadjuvant mitotane therapy will not be counted as prior drug regimens or as systemic cytotoxic chemotherapy.
* Prior radiation therapy is permitted provided patients have recovered from the acute, toxic effects of radiotherapy prior to randomization.
* A minimum of 21 days must have elapsed between the end of radiotherapy and randomization.
* Prior surgery is permitted provided that adequate wound healing has occurred prior to randomization.
* Fasting glucose < = 150 mg/dL (8.3 mmol/L).
* Adequate hematopoietic, hepatic, and renal function defined as follows: Neutrophil count >= 1.5 x 10^9 /L;
* Platelet count >= 100 x 10^9 /L;
* Bilirubin <= 1.5 x Upper Limit of Normal (ULN);
* AST and ALT <= 2.5 x ULN, or <= 5 x ULN if patient has documented liver metastases or received prior mitotane therapy; and
* Serum creatinine <= 1.5 x ULN or <= 2.0 x ULN if the patient has received prior cisplatin.
* Patients, both males and females, with reproductive potential (ie, menopausal for less than 1 year and not surgically sterilized) must agree to practice effective contraceptive measures throughout the study.
* Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to randomization.
* Patients must provide verbal and written informed consent to participate in the study.
* Radiologically-confirmed progressive disease within 6 months prior to randomization.
* Concurrent use of non-insulinotropic oral antihyperglycemic therapy is permitted if the dose has been stable for >= 4 weeks at the time of randomization.

Exclusion Criteria:

* Type 1 diabetes mellitus or Type 2 diabetes mellitus currently requiring insulinotropic or insulin therapy.
* Prior IGF-1R inhibitor therapy.
* Malignancy other than ACC within the past 3 years. Exceptions: resected basal cell or squamous cell carcinoma of the skin; cured in situ cervical carcinoma; cured ductal carcinoma in situ of the breast; and/or cured superficial bladder cancer.
* History of significant cardiovascular disease unless the disease is well-controlled.
* Significant cardiac diseases includes second/third degree heart block; clinically significant ischemic heart disease; mean QTcF interval > 450 msec at screening;
* poorly controlled hypertension; congestive heart failure of New York Heart Association (NYHA) Class II or worse (slight limitation of physical activity; comfortable at rest, but ordinary physical activity results in fatigue, palpitation, or dyspnea).
* History of cerebrovascular accident (CVA) within 6 months prior to randomization or that resulted in ongoing neurologic instability.
* Use of drugs that have a risk of causing QT interval prolongation within 14 days prior to Day 1 dosing.
* Active infection or serious underlying medical condition (including any type of active seizure disorder within 12 months prior to randomization) that would impair the ability of the patient to receive study drug.
* History of any psychiatric condition that might impair the patient's ability to understand or to comply with the requirements of the study or to provide informed consent.
* Pregnant or breast-feeding females.
* Symptomatic brain metastases that are not stable, require steroids, are potentially life threatening, or that have required radiation within 28 days prior to randomization.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2009-12-01 (Actual); Primary Completion 2012-07-11 (Actual); Study Completion 2012-10-08 (Actual)

PRIMARY OUTCOMES:
Overall survival of single agent OSI-906 versus placebo | 33 months
  Time from date of randomization until time of documented death

SECONDARY OUTCOMES:
Progression-free survival | 24 months
  Time from randomization to disease progression based on RECIST version 1.1 or death due to any cause, whichever comes first
Disease control rate | 24 months
  Proportion of patients with a best overall response of complete response (CR), partial response (PR), or stable disease (SD), based on RECIST criteria
Best overall response rate | 24 months
  Proportion of patients with a best overall response of CR or PR based on RECIST criteria
Duration of response | 24 months
  Time from date of the first documented response (CP/PR) to documented progression or death due to underlying cancer
Time to deterioration in Quality of Life | 24 months
  Measured by European Organization for the Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaires
Safety assessed via physical exams, vital signs, laboratory assessments, electrocardiograms, and adverse events | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (35):
- United States (14):
  - TGen Clinical Research Service at Scottsdale Healthcare, Scottsdale, Arizona
  - University of Southern California, Los Angeles, California
  - UCLA, Los Angeles, California
  - University of Colorado Denver Cancer Center, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - Dartmouth Medical School, Lebanon, New Hampshire
  - Duke Clinical Cancer Trials Services, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Mary Crowley Cancer Research Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Royal North Shore Hospital Department of Endocrinology, St Leonards, New South Wales, Australia
- Canada (3):
  - St. Joseph's Hospital, Hamilton, Ontario
  - PMH - Princess Margaret Hospital, Toronto, Ontario
  - Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
- France (6):
  - CHRU Lille, Clinique Endocrinologique Marc Linquette, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Hôpital Cochin-Saint Vincent de Paul, Paris
  - CHU Bordeaux - Hôpital Haut-Lévêque, Pessac
  - Institut Gustave Roussy, Villejuif
- Germany (3):
  - Charite Universitaetsmedizin, Berlin
  - LMU München, Munich
  - Universitaets Klinikum Wuerzburg, Würzburg
- Italy (2):
  - Universita di Torino, Orbassano
  - Università Cattolica del Sacro Cuore, Rome
- Netherlands (3):
  - Academic Medical Center, Amsterdam
  - Maxima Medisch Centrum (MMC), Eindhoven
  - Erasmus MC Rotterdam, Rotterdam
- Centrum Onkologii Instytut im. Marii Sklodowskiej-Curie Oddzial w Gliwicach, Gliwice, Poland
- United Kingdom (2):
  - St. James' University hospital, Leeds
  - Royal Marsden NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Fassnacht M, Berruti A, Baudin E, Demeure MJ, Gilbert J, Haak H, Kroiss M, Quinn DI, Hesseltine E, Ronchi CL, Terzolo M, Choueiri TK, Poondru S, Fleege T, Rorig R, Chen J, Stephens AW, Worden F, Hammer GD. Linsitinib (OSI-906) versus placebo for patients with locally advanced or metastatic adrenocortical carcinoma: a double-blind, randomised, phase 3 study. Lancet Oncol. 2015 Apr;16(4):426-35. doi: 10.1016/S1470-2045(15)70081-1. Epub 2015 Mar 18. PMID 25795408
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=230